CLINICAL TRIAL: NCT04956003
Title: Optimizing Cardiometabolic Health, Cognition and Academic Performance With Happy Children (HAPHC) Using School-based Physical Activity
Brief Title: Optimizing Cardiometabolic Health, Cognition and Academic Performance in Children (HAPHC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: Kristiania University College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HAPPY CHILDREN
Record Dates: First submitted 2021-06-15; First posted 2021-07-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Physical Activity; Cardiometabolic Health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention, but assessment of cardiometabolic health and cognition
- Intervention Group (Experimental): Implementing a daily 45-minute physical activity session as an integral part of learning.
  Interventions: Behavioral: 45-minute daily physical activity

INTERVENTIONS:
Behavioral: 45-minute daily physical activity — 45-minute daily physical activity session as an integral part of learning (during regular school sessions)
  Arms: Intervention Group

SUMMARY:
Children and young people are moving less and less. In combination with an unhealthy diet, this has led to a sharp increase in overweight and obesity among children worldwide. Very often, physical illnesses occur in adolescence that can be directly attributed to the overweight and obesity. In order to protect children from these consequences in time, a daily exercise unit of 45 minutes is built into their learning. This exercise will take place in addition to physical education classes as part of your child's school day and will be conducted by a teacher. We will examine the children of the participating schools with regard to health-related characteristics.

ELIGIBILITY:
Inclusion Criteria:

* students in participating schools

Exclusion Criteria:

* none

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular changes - heart rate | 3 years (4 yearly measurement time-points)
  heart rate
Cardiovascular changes - blood pressure | 3 years (4 yearly measurement time-points)
  blood pressure
Microcirculation | 3 years (4 yearly measurement time-points)
  retinal camera (retinal imaging)
Changes in subcutaneous adipose tissue | 3 years (4 yearly measurement time-points)
  Assessment via ultrasound
Changes in physical fitness - handgrip | 3 years (4 yearly measurement time-points)
  Strength via handgrip measurement
Changes in physical fitness - running | 3 years (4 yearly measurement time-points)
  Endurance via interval running test for 10 minutes
Changes in physical fitness - coordination | 3 years (4 yearly measurement time-points)
  coordination tested via Dordel-Koch-Test
Changes in cognitive performance parameters - concentration | 3 years (4 yearly measurement time-points)
  concentration tests
Changes in cognitive performance parameters - reading | 3 years (4 yearly measurement time-points)
  reading comprehension via regular school tests
Changes in cognitive performance parameters - mathematics | 3 years (4 yearly measurement time-points)
  mathematics via regular school tests

CONTACTS AND LOCATIONS:
Overall Officials: Nandu Goswami, Dr., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fredriksen PM, Hjelle OP, Mamen A, Meza TJ, Westerberg AC. The health Oriented pedagogical project (HOPP) - a controlled longitudinal school-based physical activity intervention program. BMC Public Health. 2017 Apr 28;17(1):370. doi: 10.1186/s12889-017-4282-z. PMID 28454531
- [Derived] Goswami N, Hansen D, Gumze G, Brix B, Schmid-Zalaudek K, Fredriksen PM. Health and Academic Performance With Happy Children: A Controlled Longitudinal Study Based on the HOPP Project. Front Cardiovasc Med. 2022 Jun 3;9:820827. doi: 10.3389/fcvm.2022.820827. eCollection 2022. PMID 35722126